CLINICAL TRIAL: NCT05384015
Title: A Phase II Study of Pembrolizumab, Lenvatinib and Chemotherapy Combination in First Line Extensive-stage Small Cell Lung Cancer (ES-SCLC)
Brief Title: Study of Pembrolizumab, Lenvatinib and Chemotherapy Combination in First Line Extensive-stage Small Cell Lung Cancer
Acronym: PEERS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación GECP (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GECP 20/06_PEERS; 2020-005230-15 (EudraCT Number)
Record Dates: First submitted 2022-05-17; First posted 2022-05-20 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Small Cell Lung Cancer Extensive Stage
Keywords: Lenvatinib; Pembrolizumab; Lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — lenvatinib; pembrolizumab; Etoposide; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Trial Treatment administration: at induction phase cycles will be administered every 3 weeks. For carboplatin (AUC5) and etoposide (100mg/m2) the maximum dose exposure will be 4 cycles or until reaching a discontinuation criterion. At this induction phase lenvatinib (8mg) will be orally administered daily and pembrolizumab (200mg) IV every 3 weeks. At maintenance phase lenvatinib will be administered at 20 mg dose and pembrolizumab at the same dose (200mg) until study intervention completion (total of 35 cycles of pembrolizumab/no treatment duration limit for lenvatinib) or reaching a discontinuation criterion.
  Interventions: Drug: Lenvatinib; Drug: Pembrolizumab; Drug: Etoposide; Drug: Carboplatin

INTERVENTIONS:
Drug: Lenvatinib — Lenvatinib is an oral, potent multiple receptor tyrosine kinase (RTK) i that selectively inhibits VEGF-driven VEGFR2 phosphorylation and suppressed proliferation and tube formation in human umbilical vein endothelial cell models. Antitumor activity of lenvatinib in vivo has been shown in numerous xenograft animals. These results suggest that lenvatinib may be a novel anticancer therapy through inhibition of angiogenesis and may be useful as either monotherapy or in combination with other anticancer drugs.
  Part 1 (safety run-in) and Part 2:
  The study intervention consists of:
  Dose: 8 mg (induction) and 20 mg (maintenance) Dose Frequency: Once daily Dose formulation: Capsule Route of administration: Oral Treatment duration: 4 cycles (induction) and no treatment duration limit (maintenance).
  Other Names: LENVIMA; KISPLYX
Drug: Pembrolizumab — Pembrolizumab is a potent humanized immunoglobulin G4 (IgG4) monoclonal antibody (mAb) with high specificity of binding to the programmed cell death 1 (PD-1) receptor, thus inhibiting its interaction with programmed cell death ligand 1 (PD-L1) and programmed cell death ligand 2 (PD-L2).
  Part 1 (safety run-in) and Part 2:
  Dose: 200 mg Frequency: Day 1, Q3W Route: Intravenous Treatment Period: Up to 35 cycles or until reaching a discontinuation criterion
  Other Names: KEYTRUDA
Drug: Etoposide — Standard first-line treatment for the vast majority of patients with SCLC, regardless of stage, involves combination chemotherapy with etoposide plus cisplatin or carboplatin.
  Pharmacotherapeutic group: Cytostatics, plant alkaloids and other natural products, derived from podophyllotoxin. Mechanism of action :The main effect of etoposide appears to be in the late S and early G2 phase of the cell cycle, in mammalian cells.
  Part 1 (safety run-in) and Part 2:
  Dose: 100 mg/m2 Frequency: Day 1-3, Q3W Route: Intravenous Treatment Period: 4 cycles
  Other Names: Etoposide Tevagen
Drug: Carboplatin — Pharmacotherapeutic group: Other antineoplastic agents, platinum compounds.
  Carboplatin, like cisplatin, binds to DNA to produce inter- and intra-strand cross-links cells exposed to carboplatin. DNA reactivity has been linked to cytotoxicity.
  Part 1 (safety run-in) and Part 2:
  Dose: AUC5 Frequency: Day 1, Q3W Route: Intravenous Treatment Period: 4 cycles
  Other Names: Carboplatin Accord

SUMMARY:
This is a multicenter, open-label, non-randomized, single arm, 2 parts, phase II clinical trial evaluating the efficacy and safety of pembrolizumab and lenvatinib plus standard of care chemotherapy (with carboplatin and etoposide ) in subjects with histologically confirmed extensive-stage small-cell lung cancer who have not previously received systemic therapy for this malignancy.

DETAILED DESCRIPTION:
A total of 85 subjects will be assigned to study treatment with pembrolizumab + lenvatinib + chemotherapy. Positive tumor programmed cell death-ligand 1 (PD-L1) expression will not be required for enrollment; however, subjects' tumors will be screened for PD-L1 expression.

The primary endpoint for the Part 1 is to determine the safety of the combination. The primary endpoint for Part 2 is to determine the Progression Free survival (PFS) using RECIST 1.1. assessed by investigator.

The sponsor estimates that the trial will require approximately 4 years from the time the first participant signs the informed consent until the last participant's last study-related telephone call or visit (2 years recruiting patients, 1 year of treatment and at least 1 year of follow up)

ELIGIBILITY:
Inclusion Criteria:

- 1. Histologically or cytologically documented new diagnosis of SCLC by histology or cytology from brushing, washing, or needle aspiration.

Note: Subjects who do not have histology samples (defined as core or excisional biopsy, or resections) will need to undergo a new biopsy to provide a tissue sample. Mixed tumors are not eligible.

* 2. ES-SCLC, stage IV disease by the American Joint Committee on Cancer, 8th Edition criteria (70), [T any, N any, M1a, M1b, M1c], or T3-4 due to multiple lung nodules that are too extensive or tumor/nodal volume that is too large to be encompassed in a tolerable radiation plan.
* 3. Have at least one lesion that meets criteria for being measurable, as defined by RECIST 1.1.
* 4. Have provided archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated for biomarker assessment.
* 5. Be male or female ≥18 years of age inclusive, on the day of signing informed consent.
* 6. Have a life expectancy of at least 3 months from the study start.
* 7. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 within 7 days prior to the first dose of study intervention.
* 8. Male participants are eligible to participate if they agree to the following during the intervention period and for at least 30 days after the last dose of lenvatinib placebo and up to 180 days after the last dose of chemotherapeutic agents:

  * Refrain from donating sperm

PLUS either:

* Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent OR
* Must agree to use contraception unless confirmed to be azoospermic.

  - 9. A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:
* Is not a WOCBP OR
* Is a WOCBP and using a contraceptive method that is highly effective

  * 10. Have voluntarily agreed to participate by giving written consent for the study prior to any specific protocol procedures.
  * 11. Have adequate organ function

Exclusion Criteria:

* 1. Has received any prior therapy (chemotherapy, radiotherapy, surgical resection) or other investigational agent for the treatment of SCLC.
* 2. Is expected to require any other form of antineoplastic therapy for SCLC, including radiation therapy while on study.
* 3. Active CNS metastases and/or carcinomatous meningitis as determined per CT or MRI during screening. Participants with previously treated brain metastases (eg, whole brain radiation treatment [WBRT], stereotactic radiosurgery, or equivalent) may participate only if they satisfy the following:

  * Completed treatment at least 14 days prior to the first dose of study intervention.
  * Are clinically stable, without requirement of steroid treatment for at least 7 days prior to first dose of study intervention.
  * Are radiologically stable.
  * Patients with new asymptomatic CNS metastases detected at the screening scan must receive radiation therapy and/or surgery for CNS metastases. Following treatment, these patients may then be eligible without the need for an additional brain scan prior to enrollment, if all other criteria are met.
* 4. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137).
* 5. Spinal cord compression not definitively treated with surgery and/or radiation or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for ≥ 1 week prior to enrollment.
* 6. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently). A subject who is clinically stable following treatment for these conditions (including therapeutic thoraco- or paracentesis) is eligible.
* 7. .Has known history of, or active, neurologic paraneoplastic syndrome of autoimmune nature.
* 8. Radiographic evidence of intratumoral cavitations, encasement, or invasion of a major blood vessel. Additionally, the degree of proximity to major blood vessels should be considered for exclusion because of the potential risk of severe hemorrhage associated with tumor shrinkage/necrosis after lenvatinib therapy.
* 9. Has had major surgery within 4 weeks prior to first dose of study interventions.
* 10. Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of trial drug.
* 11. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.
* 12. Has an active autoimmune disease or inflammatory disorder that has required systemic treatment in the past 2 years.
* 13. Has a diagnosis of immunodeficiency or is taking chronic systemic steroid therapy (in dosing of >10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* 14. Has known history of a second malignancy other than SCLC, unless potentially curative treatment has been completed with no evidence of malignancy for at least 3 years since the initiation of that therapy.
* 15. Poor controlled hypertension (BP>150/90 mmHg) despite appropriate treatment.
* 16. Participants with proteinuria >1+ on urine dipstick testing/urinalysis will undergo 24-hour urine collection for quantitative assessment of proteinuria. Participants with urine protein ≥1 g/24 hours will be ineligible.
* 17. Has a prolongation of QTc interval (calculated using Fridericia's formula) of >480 msec.
* 18. Has a known history of interstitial lung disease, idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan
* 19. Uncontrolled intercurrent active infection at the time of enrollment requiring systemic therapy.
* 20. Has a known history of Human Immunodeficiency Virus (HIV) infection.
* 21. Has a known history of Hepatitis B or known active Hepatitis C.
* 22. Has a known history of active tuberculosis.
* 23. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study.
* 24. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* 25. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study.
* 26. Prior allogeneic bone marrow transplantation or solid organ transplant.
* 27. Any gastrointestinal condition that would affect the absorption of Lenvatinib.
* 28. Has active hemoptysis or major arterial thromboembolic event within 2 weeks prior to the first dose of study intervention.
* 29. Has significant cardiovascular impairment within 12 months prior to the first dose of study intervention.
* 30. Has a history of a severe (Grade ≥ 3) hypersensitivity reaction to treatment with another monoclonal antibody or has a known hypersensitivity to lenvatinib, pembrolizumab, carboplatin or etoposide and/or any of its excipients.
* 31. Has a clinically active diverticulitis, inflammatory bowel disease, intra-abdominal abscess, gastrointestinal obstruction and/or abdominal carcinomatosis.
* 32. Has a history of a gastrointestinal perforation within 6 months before the first dose of study intervention.
* 33. Has preexisting Grade ≥ 3 gastrointestinal or non-gastrointestinal fistula.
* 34. Has serious nonhealing wound, ulcer, or bone fracture within 28 days before first dose of study intervention.
* 35. Has any major hemorrhage or venous thromboembolic events within 3 months before the first dose of study intervention.
* 36. Poor medical risk due to a serious, uncontrolled medical disorder or nonmalignant systemic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2022-11-07 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Part 1: Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) of lenvatinib 8 mg to be used in combination with pembrolizumab plus chemotherapy | From the subject's written consent to participate in the study through 90 days after the final administration of the drug
  Occurrence and severity of adverse events, with severity determined by NCI CTCAE v5.0 criteria.
Part 2:To assess the efficacy of the treatment in terms of the Progression Free Survival (PFS) | From the date of the end of induction treatment until 12 months
  PFS is defined as the time from enrollment to the date of the first documentation of disease progression, as determined by investigator per RECIST 1.1, or death from any cause, whichever is earlier.

SECONDARY OUTCOMES:
Part 1 (for patients treated at part 2): Objective response per RECIST 1.1 based on investigator | From the date of the end of treatment until 12 months
  Objective response is a confirmed complete response (CR) or partial response (PR), as determined by investigator per RECIST 1.1.
Part 1 (for patients treated at part 2): Duration of Response (DOR) per RECIST 1.1 based on investigator | From date of documentation of tumor response until date of first documented progression, assessed up to 12 months
  DOR is defined as the time from the first documented evidence of CR or PR until disease progression or death due to any cause (whichever is earlier), for participants who demonstrate a confirmed CR or PR. Response will be determined by BICR per RECIST 1.1.
Part 1 (for patients treated at part 2): Overall Survival | From the date of the end of treatment until 12 months
  OS is defined as the time from enrollment to the date of death from any cause.
Part 2: Objective response per RECIST 1.1 based on investigator | From the date of the end of treatment until 12 months
  Objective response is a confirmed complete response (CR) or partial response (PR), as determined by investigator per RECIST 1.1.
Part 2: Duration of Response (DOR) per RECIST 1.1 based on investigator | From date of documentation of tumor response until date of first documented progression, assessed up to 12 months
  DOR is defined as the time from the first documented evidence of CR or PR until disease progression or death due to any cause (whichever is earlier), for participants who demonstrate a confirmed CR or PR. Response will be determined by BICR per RECIST 1.1.
Part 2:Overall Survival | From the date of the end of treatment until 12 months
  OS is defined as the time from enrollment to the date of death from any cause.
Part 2: Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) of treatment | From the subject's written consent to participate in the study through 90 days after the final administration of the drug
  Occurrence and severity of adverse events, with severity determined by NCI CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Noemí Reguart, MD, Study Chair — Principal Investigator of Fundación Grupo Español de Cáncer de Pulmón
Locations (18):
- Spain (18):
  - ICO Badalona, Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospitalario Universitario A Coruña, A Coruña, La Coruña
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitari Vall d' Hebron, Barcelona
  - Hospital Clínic De Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Parc Taulí, Barcelona
  - Hospital De Basurto, Bilbao
  - ICO Girona, Hospital Josep Trueta, Girona
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital 12 De Octubre, Madrid
  - Hospital Universitario Regional de Málaga, Málaga
  - Hospital Son Espases, Palma de Mallorca
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Clínico de Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Description Web page of the sponsor where users can find more information about Fundacion GECP studies. — http://www.gecp.org